CLINICAL TRIAL: NCT05646186
Title: Comparison of Personalized Diet Implementation Based on Microbiome Analysis and FODMAP Diet Efficacy in Irritable Bowel Syndrome
Brief Title: Personalized Dietary Intervention Based on Microbiome Analysis vs FODMAP Diet for Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Bozyaka Training and Research Hospital (Other); Tepecik Training and Research Hospital (Other); Dr. Ersin Arslan Education and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E-10840098-772.02-5763
Record Dates: First submitted 2022-10-06; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-09

CONDITIONS: Irritable Bowel Syndrome; Irritable Bowel Syndrome With Diarrhea; Irritable Bowel Syndrome With Constipation; Irritable Bowel Syndrome Mixed
Keywords: Microbiome; Microbiota; Personalised medicine; Artificial intelligence
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blinded randomized controlled study. The participants will be blinded to the dietary interventions and the care providers will apply the diets that were allocated to them without knowing which diet they are applying. The investigators will not be able to obtain data until the data collection is finished.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalised diet based on microbiome analysis (Experimental): Personalized diet application based on artificial intelligence-assisted microbiome analysis. After the microbiome analysis is made from the stool samples to be taken from the individuals, a personalized diet program will be created with an artificial intelligence-based algorithm and a diet will be applied for 6 weeks with the support of a professional dietitian.
  Interventions: Dietary Supplement: Personalized dietary intervention based on microbiome analysis
- Low FODMAP diet (Active Comparator): After the microbiome analysis is made from the stool samples to be taken from the individuals, low fermentable oligosaccharides, disaccharides, monosaccharides, and polyols (FODMAP) diet will be applied for 6 weeks with the support of a professional dietitian.
  Interventions: Dietary Supplement: Low-FODMAP diet

INTERVENTIONS:
Dietary Supplement: Personalized dietary intervention based on microbiome analysis — Personalized dietary intervention based on individual microbiome analysis
  Other Names: Enbiosis IBS Scheme
  Arms: Personalised diet based on microbiome analysis
Dietary Supplement: Low-FODMAP diet — Low fermentable oligosaccharides, disaccharides, monosaccharides, and polyols diet
  Arms: Low FODMAP diet

SUMMARY:
irritable bowel syndrome (IBS) is a well-known risk factor for diseases of the anal region (hemorrhoids, anal fissures, etc.) and large intestine (colon cancer, diverticular disease). Untreatable IBS disease not only impairs the patient's quality of life but also reduces the success of surgical treatment in these diseases.

Today, only one-third of IBS patients achieve successful results with the treatment methods and diets used routinely. Balancing the composition of the gut microbiota may yield satisfactory results in this patient group. With the results of our study, we aim to reveal the effect of microbiome analysis and personalized diet on symptoms and its place in treatment in patients with IBS disease.

Patients applying to Gastroenterology outpatient clinics in respective centers due to IBS will be randomized into two groups. The patients in the control group will follow the FODMAP diet protocol for IBS; In the study group, a personalized diet will be applied according to the gut microbiota. No nutritional supplements will be used in either group. Changes in defecation habits and quality of life scale of both groups will be evaluated at the end of 6 weeks and the results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-65
* To be diagnosed with IBS (IBS-D, IBS-C, IBS-M) according to the Rome IV Criteria
* To give consent to participate in the study voluntarily
* Being a smartphone and/or internet user (for dietitian follow-up and clinical follow-up)
* Not meeting any of the exclusion criteria

Exclusion Criteria:

* Pregnant or planning to become pregnant
* Having another known diagnosis of gastrointestinal disease (inflammatory bowel disease, malabsorption of any macronutrient, intestinal resection, celiac disease, etc.)
* Colonoscopy history (in the last 1 year)
* History of abdominal surgery other than appendectomy or hysterectomy
* Psychiatric comorbidity
* Chronic diseases that will affect the microbiome (cancer, diabetes, cardiovascular disease, liver diseases, neurological diseases, etc.)
* Use of drugs that may affect digestive function in the 4 weeks prior to the study (antibiotics (including use in the last 4 weeks), probiotics, narcotic analgesics, lactulose (prebiotics))
* Patients taking dietary supplements
* Excluded from the study if following a restricted diet.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in IBS Symptom severity score | 6 weeks
  Change in IBS Symptom severity score after 6 weeks of dietary intervention
Change in IBS quality of life scale | 6 weeks
  Change in IBS quality of life scale after 6 weeks of dietary intervention
Change in Anxiety-depression scale | 6 weeks
  Change in Anxiety and depression scale after 6 weeks of dietary intervention

SECONDARY OUTCOMES:
Difference between study and control arms | 6 months
  A statistically significant difference between study and control groups based on the IBS-SSS, IBS-QOL and Anxiety depression scale

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University Bahcelievler Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be made available in a data repository

REFERENCES:
- [Derived] Tunali V, Arslan NC, Ermis BH, Dervis Hakim G, Gundogdu A, Hora M, Nalbantoglu OU. A Multicenter Randomized Controlled Trial of Microbiome-Based Artificial Intelligence-Assisted Personalized Diet vs Low-Fermentable Oligosaccharides, Disaccharides, Monosaccharides, and Polyols Diet: A Novel Approach for the Management of Irritable Bowel Syndrome. Am J Gastroenterol. 2024 Sep 1;119(9):1901-1912. doi: 10.14309/ajg.0000000000002862. Epub 2024 May 8. PMID 38717025